CLINICAL TRIAL: NCT01738217
Title: Evaluation, for Patients Requiring a Liver Cancer Surgery, of the Use of Fluorescence Imaging Device: Faisability and Efficiency of Lesional and/or Anatomical Marking
Brief Title: Assessment of Indocyanine Green as a Near-Infrared Fluorescent Contrast Agent for Image-guided Liver Surgery
Acronym: HEPATOFLUO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HEPATOFLUO; ET12-066 (Other: Sponsor Number)
Record Dates: First submitted 2012-11-26; First posted 2012-11-30 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Liver Neoplasms
Keywords: Intra-operative imaging; NIR Fluorescence; Liver surgery; Tumoral margins
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fluobeam (Experimental)
  Interventions: Procedure: Fluobeam

INTERVENTIONS:
Procedure: Fluobeam

SUMMARY:
This is a prospective, monocentric, non-randomized, phase I-II study. The goal is to assess the faisability and the capabilities of fluorescence imaging in hepatic surgery, and specially to help the surgeon while performing liver surgery.

This study will be performed on patient intended to undergo a liver cancer surgery.It will contain three steps, assessing the following items:

* Step 1: to assess the faisability of the use of the Fluobeam, in actual clinical surgical conditions and validate the data obtained in the preclinical phase,
* Step 2: to assess the ability of the combination of ICG and Fluobeam to mark hepatic lesions,
* Step 3: to assess the ability of the combination of ICG and Fluobeam to help in guiding per-hepatectomy.

  3 to 6 patients will be enrolled in the first step, 20 in the second step and 20 in the third step.

Patients will be followed during 4 weeks after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Affected of hepatic cancerous lesions whatever they are
* Requiring a one or two steps hepatectomy by laparotomy
* ECOG performance status (PS)≤ 2
* Mandatory affiliation to health security insurance
* Written informed consent

Exclusion Criteria:

* With a contraindication or hypersensitivity to ICG administration in medical history
* Having already undergone a major hepatic surgery (more than three segments) or major biliar surgery (context of major iterative hepatic surgery)
* Unable to be followed during the duration of the study, for social, family, geographical or psychological reasons
* Pregnant or breast-feeding woman (urinary strip must be negative at the time of the inclusion in the study for women in age to procreate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
First step: assess the feasibility and the acceptability of Fluobeam | During surgery on day 0
  * The ability to detect fluorescence
  * The ability to investigate the mobilized parenchyma
  * The ability to use the medical device following requested asepsis procedures
  * Surgeon satisfaction
  * Nurse satisfaction
Second step: assess the rate of patients in whom, all of the lesions (superficial/deep) will be detected by means of the Fluobeam medical device in peroperative or in postoperative. | During surgery on day 0
Third step: assess the rate of patients in whom, among the 7 liver segments, the surgeon will be able to selectively target a predefined area. | During surgery on day 0

SECONDARY OUTCOMES:
First step: assess the ability to visualize the fluorescent anatomical areas | During surgery on day 0
First step: Quantify the fluorescence | After the surgery, on day 0
  by using the images obtained during the surgery
First step: assess the ability to review saved data | After the surgery, on day 0
Second step: assess the ability to detect tumor lesions which were not previously known. | During surgery on day 0
  Assessment of the number of lesions detected thanks to the medical device. The malignant aspect must be confirmed by an anatomopathological analysis.
Second step: assess the rate of modifications of the surgical plan. | During surgery on day 0
  Number of patients for whom the surgery would be modified after using Fluobeam.
Second step: assess the quality of the resection margins. | After the surgery on day 0
  It will be measured using the residual fluorescence and the pathology analysis
Second step: assess the depth limit of detection of the fluorescence. | After the pathology analysis on day 0
  It will be assessed after the anatomopathological analysis.
Second step: Quantify the fluorescence. | After the surgery, on day 0
  From images obtained during the surgery and from the sample analysed by a pathologist.
Second step: assess the number of asepsis due to Fluobeam | During surgery on day 0
Third step: assess the ability to detect tumor lesions which were not previously known. | During surgery on day 0
  Assessment of the number of lesions detected thanks to the medical device. The malignant aspect must be confirmed by an anatomopathological analysis
Third step: quantify the fluorescence. | After the surgery on day 0
  From images obtained during the surgery and from the sample analysed by a pathologist.
Third step: assess the ability to administer two doses of ICG in the same patient | On day 0
  one before and one during the surgery (tumor detection and segment targeting respectively).
Third step: assess the number of asepsis due to Fluobeam | During surgery on day 0
Third step: assess the ability of the medical device to detect tumor lesions which were previously known. | On day 0
  Number of lesions seen on images before and during the surgery and detected by Fluobeam.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Peyrat, Principal Investigator — Centre Léon Bérard, LYON, FRANCE.
Locations (1):
- Centre Léon Bérard, Lyon, France

REFERENCES:
- [Background] Aoki T, Murakami M, Yasuda D, Shimizu Y, Kusano T, Matsuda K, Niiya T, Kato H, Murai N, Otsuka K, Kusano M, Kato T. Intraoperative fluorescent imaging using indocyanine green for liver mapping and cholangiography. J Hepatobiliary Pancreat Sci. 2010 Sep;17(5):590-4. doi: 10.1007/s00534-009-0197-0. Epub 2009 Oct 21. PMID 19844652
- [Background] Aoki T, Yasuda D, Shimizu Y, Odaira M, Niiya T, Kusano T, Mitamura K, Hayashi K, Murai N, Koizumi T, Kato H, Enami Y, Miwa M, Kusano M. Image-guided liver mapping using fluorescence navigation system with indocyanine green for anatomical hepatic resection. World J Surg. 2008 Aug;32(8):1763-7. doi: 10.1007/s00268-008-9620-y. PMID 18543027
- [Background] Barbare JC. Quantification de la fonction hépatique: Pourquoi et comment? John Libbey Eurotext. HEPATO-GASTRO.5(6):423-431,1998.
- [Background] Billingsley KG, Jarnagin WR, Fong Y, Blumgart LH. Segment-oriented hepatic resection in the management of malignant neoplasms of the liver. J Am Coll Surg. 1998 Nov;187(5):471-81. doi: 10.1016/s1072-7515(98)00231-2. PMID 9809562
- [Background] Gotoh K, Yamada T, Ishikawa O, Takahashi H, Eguchi H, Yano M, Ohigashi H, Tomita Y, Miyamoto Y, Imaoka S. A novel image-guided surgery of hepatocellular carcinoma by indocyanine green fluorescence imaging navigation. J Surg Oncol. 2009 Jul 1;100(1):75-9. doi: 10.1002/jso.21272. PMID 19301311
- [Background] Hamamatsu Photonics-Pulsion Medical System.PDE Photodynamic Eye. http://www.iht-ltd.com/pde-photodynamic-eye/
- [Background] Hamoui M; Marchand JP. Boutabrine H. Navarro F. L'évaluation préopératoire du risque d'insuffisance hépatocellulaire lors des résections hépatiques sur foie cirrhotique. John Libbey Eurotext.HEPATO-GASTRO. 16(1):11-19, 2009
- [Background] HAS.Guide ALD30-Tumeur maligne, affection maligne du tissu lymphatique ou hématopoïétique-Cancer primitif du foie. http://www.e-cancer.fr/soins/recommandations/cancers-digestifs
- [Background] HAS. Guide ALD-Tumeur maligne, affection maligne du tissu lymphatique ou hématopoïétique-Cancer colorectal Adénocarcinome. http://www.e-cancer.fr/soins/recommandations/cancers-digestifs
- [Background] Ishizawa T, Fukushima N, Shibahara J, Masuda K, Tamura S, Aoki T, Hasegawa K, Beck Y, Fukayama M, Kokudo N. Real-time identification of liver cancers by using indocyanine green fluorescent imaging. Cancer. 2009 Jun 1;115(11):2491-504. doi: 10.1002/cncr.24291. PMID 19326450
- [Background] Ishizuka M, Kubota K, Kita J, Shimoda M, Kato M, Sawada T. Intraoperative observation using a fluorescence imaging instrument during hepatic resection for liver metastasis from colorectal cancer. Hepatogastroenterology. 2012 Jan-Feb;59(113):90-2. doi: 10.5754/hge11223. PMID 22260827
- [Background] Jarnagin WR, Bach AM, Winston CB, Hann LE, Heffernan N, Loumeau T, DeMatteo RP, Fong Y, Blumgart LH. What is the yield of intraoperative ultrasonography during partial hepatectomy for malignant disease? J Am Coll Surg. 2001 May;192(5):577-83. doi: 10.1016/s1072-7515(01)00794-3. PMID 11333094
- [Background] Morita Y, Sakaguchi T, Unno N, Shibasaki Y, Suzuki A, Fukumoto K, Inaba K, Baba S, Takehara Y, Suzuki S, Konno H. Detection of hepatocellular carcinomas with near-infrared fluorescence imaging using indocyanine green: its usefulness and limitation. Int J Clin Oncol. 2013 Apr;18(2):232-41. doi: 10.1007/s10147-011-0367-3. Epub 2011 Dec 27. PMID 22200990
- [Background] O2View. ArteMIS Handheld Complete System. http://o2view.com/
- [Background] Pawlik TM, Scoggins CR, Zorzi D, Abdalla EK, Andres A, Eng C, Curley SA, Loyer EM, Muratore A, Mentha G, Capussotti L, Vauthey JN. Effect of surgical margin status on survival and site of recurrence after hepatic resection for colorectal metastases. Ann Surg. 2005 May;241(5):715-22, discussion 722-4. doi: 10.1097/01.sla.0000160703.75808.7d. PMID 15849507
- [Background] Reuthebuch O, Haussler A, Genoni M, Tavakoli R, Odavic D, Kadner A, Turina M. Novadaq SPY: intraoperative quality assessment in off-pump coronary artery bypass grafting. Chest. 2004 Feb;125(2):418-24. doi: 10.1378/chest.125.2.418. PMID 14769718
- [Background] Rivoire M.Diagnostiquer une tumeur du foie primitive et secondaire. http://cancero.unice.fr/sitelocal/disciplines/niveaudiscipline/cancerologie/numlecon151/leconimprim.pdf
- [Background] Schaafsma BE, Mieog JS, Hutteman M, van der Vorst JR, Kuppen PJ, Lowik CW, Frangioni JV, van de Velde CJ, Vahrmeijer AL. The clinical use of indocyanine green as a near-infrared fluorescent contrast agent for image-guided oncologic surgery. J Surg Oncol. 2011 Sep 1;104(3):323-32. doi: 10.1002/jso.21943. Epub 2011 Apr 14. PMID 21495033
- [Background] Société Française de Chirurgie Digestive (SFCD), Association de Chirurgie hépatobiliaire et de Transplantation Hépatique (ACHBT). Prise en charge des patients atteints de métastases hépatiques synchrones du cancer colorectal-Recommandations professionnelles-Synthèse. www.e-cancer.fr
- [Background] Takahashi M, Ishikawa T, Higashidani K, Katoh H. SPY: an innovative intra-operative imaging system to evaluate graft patency during off-pump coronary artery bypass grafting. Interact Cardiovasc Thorac Surg. 2004 Sep;3(3):479-83. doi: 10.1016/j.icvts.2004.01.018. PMID 17670291
- [Background] Weber SM, Jarnagin WR, DeMatteo RP, Blumgart LH, Fong Y. Survival after resection of multiple hepatic colorectal metastases. Ann Surg Oncol. 2000 Oct;7(9):643-50. doi: 10.1007/s10434-000-0643-3. PMID 11034240
- [Result] Slim K, Blay JY, Brouquet A, Chatelain D, Comy M, Delpero JR, Denet C, Elias D, Flejou JF, Fourquier P, Fuks D, Glehen O, Karoui M, Kohneh-Shahri N, Lesurtel M, Mariette C, Mauvais F, Nicolet J, Perniceni T, Piessen G, Regimbeau JM, Rouanet P, sauvanet A, Schmitt G, Vons C, Lasser P, Belghiti J, Berdah S, Champault G, Chiche L, Chipponi J, Chollet P, De Baere T, Dechelotte P, Garcier JM, Gayet B, Gouillat C, Kianmanesh R, Laurent C, Meyer C, Millat B, Msika S, Nordlinger B, Paraf F, Partensky C, Peschaud F, Pocard M, Sastre B, Scoazec JY, Scotte M, Triboulet JP, Trillaud H, Valleur P. [Digestive oncology: surgical practices]. J Chir (Paris). 2009 May;146 Suppl 2:S11-80. doi: 10.1016/S0021-7697(09)72398-1. No abstract available. French. PMID 19435621